CLINICAL TRIAL: NCT05396391
Title: A Phase I/IIa Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Effectiveness of IAP0971 in Patients With Advanced Malignant Tumors
Brief Title: A Clinical Trial to Evaluate Effect of IAP0971 in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IAP0971-I/IIa
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Advanced Malignant Tumors
Keywords: PD1; IL15; Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase Ia - Dose escalation (Experimental): The goal of the Dose Escalation Phase (Part A) is to initially characterize the safety and tolerability of IAP0971, and more specifically to describe the DLTs for each dose level studied and to define the MTD based on the frequency of the occurrence of DLTs in each cohort during the DLT evaluation period.
  Interventions: Drug: IAP0971
- Phase Ib - Dose extension (Experimental): During the Dose Expansion Phase , patients will be enrolled to receive IAP0971 at the MTD established from the Dose Escalation Phase of the study.
  Interventions: Drug: IAP0971
- Phase IIa - Clinical Exploratory Stage (Experimental): After finishing Phase 1, invesigators will discuss with the sponsor about how to carry out the Phase IIa due to the results acheived from Phase I.
  Interventions: Drug: IAP0971

INTERVENTIONS:
Drug: IAP0971 — IAP0971 should be subcutaneous injected，q2w

SUMMARY:
This is a Phase I Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Effectiveness of IAP0971 in Patients with Advanced Malignant Tumors.

DETAILED DESCRIPTION:
The study includes three phases: dose escalation (Phase Ia), dose extension (Phase Ib), and clinical exploration (Phase IIa).First, the Phase Ia dose escalation will be carried out. After finishing the Phase 1a，the Phase Ib dose extension study can be carried out in the MTD dose which can be achieved from Phase 1a. After Phase Ia & Ib are completed and RP2D is obtained, Phase IIa clinical exploratory research can be carried out.

ELIGIBILITY:
Inclusion Criteria:

- 1. Age 18 to 80 years, male or female. 2. Patients with histologically or cytologically confirmed advanced or unresectable solid tumors or and relapsed and/or refractory non-Hodgkin's lymphoma, who have progressed on or have been intolerant to standard treatment, or for whom no standard treatment exists.

3. Dose Escalation Phase (Part A)：At least one evaluable tumor lesion per RECIST 1.1 (solid tumors) or Lugano 2014 (lymphomas).

Dose Expansion Phase (Part B)：At least one measurable tumor lesion per RECIST 1.1 (solid tumors) or Lugano 2014 (lymphomas).

4. Agree to provide previously stored tumor tissue specimens or perform biopsy to collect tumor lesion tissue and send it to the central laboratory for PD-L1 expression level detection.

5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. (see Appendix 3) 6. Adequate organ function: Hematological system (No blood transfusion or hematopoietic stimulating factor therapy within 14 days) Absolute neutrophil count (ANC) ≥ 1.5 × 109/L White blood cell count (WBC) ≥ 3.0 × 109/L Platelets (PLT) ≥ 75 × 109/L Hemoglobin (Hb) ≥ 90 g/L Hepatic function Total bilirubin (TBIL) ≤ 3 × ULN Alanine aminotransferase (ALT) ≤ 3 × ULN; Aspartate aminotransferase (AST) ≤ 3 × ULN; Renal function Creatinine clearance (Ccr) (only calculated if creatinine > 3 × ULN) ≥ 50 mL/min (calculated according to Cockcroft-Gault formula, see Appendix 7 for formula) Coagulation function Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN International normalized ratio (INR) ≤ 1.5 × ULN 7. Expected survival time of more than 3 months. 8. Eligible patients of childbearing potential (men and women) must agree to use a reliable method of contraception (hormonal or barrier method or abstinence, etc.) with their partners during the trial and for at least 90 days after study drug administration; female patients of childbearing potential (see Appendix 8 for definition) must have a negative blood or urine pregnancy test 7 days before the first administration.

9. Subjects must be informed of the study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

- 1. Patients who have a severe hypersensitivity reaction to any monoclonal antibody (CTCAE 5.0 grade ≥ 3).

2. Patients who received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, and other anti-tumor treatment within 4 weeks before the first administration, except for the following: Nitrosourea or mitomycin C was received within 6 weeks before the first administration; Oral fluoropyrimidines and small molecule targeted drugs within 2 weeks or 5 half-lives of the drug (whichever is longer) prior to the first administration.

Chinese proprietary medicines with anti-tumor indications were received within 2 weeks before the first administration.

3. Receipt of other non-marketed investigational drugs or treatments within 4 weeks before the first administration.

4. Patients who have undergone major organ surgery (excluding needle biopsy) or have significant trauma within 4 weeks before the first administration, or require elective surgery during the trial.

5. Patients who have received systemic glucocorticoids (prednisone > 10 mg/day or equivalent doses of similar drugs) or other immunosuppressive agents within 14 days before the first administration; exclude the following conditions: topical, ophthalmic, intra-articular, intranasal or inhaled corticosteroid therapy; short-term use of glucocorticoid for preventive treatment (for example, prevention of contrast agent allergy).

6. Patients who have received immunomodulatory drugs within 14 days before the first administration, including but not limited to thymosin, interleukin-2, interferon, etc.

7. Patients who have received live attenuated vaccines within 4 weeks before the first administration.

8. Previous allogeneic hematopoietic stem cell transplantation or organ transplantation.

9. The adverse reactions caused by previous anti-tumor treatment have not recovered to CTCAE 5.0 grade ≤ 1 (except for toxicity without safety risk as judged by the investigator, such as alopecia, grade 2 peripheral neurotoxicity, hypothyroidism stabilized by hormone replacement therapy, etc.).

10. Patients with active infection who need intravenous anti-infective therapy. 11. Patients with interstitial lung disease (except for radiation pulmonary fibrosis not requiring hormone therapy).

12. History of serious cardiovascular and cerebrovascular diseases, including but not limited to: Patients with severe cardiac rhythm or conduction abnormalities, such as arrhythmia requiring clinical intervention, second-degree to third-degree atrioventricular block; QT interval (QTcF) corrected by Fridericia's method > 470 ms (see Appendix 9 for calculation formula); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 and above cardiovascular and cerebrovascular events within 6 months prior to the first dose; Patients with heart failure with cardiac function class ≥ II according to New York Heart Association (NYHA) (see Appendix 4) or Left Ventricular Ejection Fraction (LVEF) < 50%; Clinically uncontrolled hypertension. 13. Patients who currently have active or have had autoimmune diseases that may have recurrence (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for clinically stable autoimmune thyroid diseases, type I Diabetics.

14. Patients who have received immunotherapy and developed irAE ≥3 or immune-related myocarditis ≥2.

15. Clinically uncontrolled effusion in the third space, which is not suitable for enrollment based on the investigator's judgment.

16. Known alcohol or drug dependence. 17. Patients with mental disorders or poor compliance. 18. Women who are pregnant or breastfeeding. 19. The subject has a history of other serious systemic diseases or other reasons that make the subject unsuitable for this clinical study in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of IAP0971 (Phase I) | Through finishing Phase I, an average of 1 year
  MTD/RP2D; Incidence and frequency of DLT; AE, SAE occurrence and frequency (according to NCI CTCAE 5.0).
To evaluate the effectiveness of IAP0971 (Phase IIa) | Until disease progression, assessed up to 3 years
  Objective response rate(ORR)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) Cmax（Phase I) | After single dose ,assessed up to 1 year
  PK parameters Cmax following single dose
Pharmacokinetics (PK) Css,max（Phase I) | After multiple doses ,assessed up to 1 year
  PK parameters Css,max following multiple doses
Pharmacokinetics (PK) Css,min（Phase I) | After multiple doses ,assessed up to 1 year
  PK parameters Css,min following multiple doses
Pharmacokinetics (PK) Css,av（Phase I) | After multiple doses ,assessed up to 1 year
  PK parameters Css,av following multiple doses
Pharmacokinetics (PK) AUCss（Phase I) | After multiple doses ,assessed up to 1 year
  PK parameters AUCss following multiple doses
Pharmacokinetics (PK) CLss（Phase I) | After multiple doses ,assessed up to 1 year
  PK parameters CLss following multiple doses
Pharmacokinetics (PK) Vss（Phase I) | After multiple doses ,assessed up to 1 year
  PK parameters Vss following multiple doses
Pharmacokinetics (PK) R（Phase I) | After multiple doses ,assessed up to 1 year
  PK parameters R following multiple doses
Pharmacokinetics (PK) DF（Phase I) | After multiple doses ,assessed up to 1 year
  PK parameters DF following multiple doses
Pharmacokinetics (PK) Tmax（Phase I) | After single dose ,assessed up to 1 year
  PK parameters Tmax following single dose
Pharmacokinetics (PK) AUC0-t（Phase I) | After single dose ,assessed up to 1 year
  PK parameters AUC0-t following single dose
Pharmacokinetics (PK) AUC0-∞（Phase I) | After single dose ,assessed up to 1 year
  PK parameters AUC0-∞ following single dose
Pharmacokinetics (PK) CL（Phase I) | After single dose ,assessed up to 1 year
  PK parameters CL following single dose
Pharmacokinetics (PK) Vd（Phase I) | After single dose ,assessed up to 1 year
  PK parameters Vd following single dose
Pharmacokinetics (PK) t1/2（Phase I) | After single dose ,assessed up to 1 year
  PK parameters t1/2 following single dose
Pharmacokinetics (PK) λz（Phase I) | After single dose ,assessed up to 1 year
  PK parameters λz following single dose
To evaluate the immunogenicity of IAP0971 in patients with advanced malignant tumors (Phase I) | After finishing Phase I, an average of 1 year
  Incidence of anti-drug antibody (ADA) and neutralizing antibodies (NAb) against IAP0971
To evaluate the effectiveness of IAP0971 in patients with advanced malignant tumors (Phase I) | After finishing Phase I, an average of 1 year
  Overall survival (OS) according to RECIST 1.1 or Lugano 2014
To evaluate the effectiveness of IAP0971 in patients with advanced malignant tumors (Phase I) | After finishing Phase I, an average of 1 year
  Objective response rate (ORR) according to RECIST 1.1 or Lugano 2014
To evaluate the immunogenicity of IAP0971 in patients with advanced malignant tumors (Phase IIa) | After finishing Phase IIa, assessed up to 3 years
  Incidence of anti-drug antibody (ADA) and neutralizing antibodies (NAb) against IAP0971
o evaluate the effectiveness of IAP0971 in patients with advanced malignant tumors (Phase IIa) | After finishing Phase IIa, assessed up to 3 years
  PFS according to RECIST 1.1 or Lugano 2014
o evaluate the effectiveness of IAP0971 in patients with advanced malignant tumors (Phase IIa) | After finishing Phase IIa, assessed up to 3 years
  DCR according to RECIST 1.1 or Lugano 2014
o evaluate the effectiveness of IAP0971 in patients with advanced malignant tumors (Phase IIa) | After finishing Phase IIa, assessed up to 3 years
  OS according to RECIST 1.1 or Lugano 2014

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D., Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Shen Z, Jiang X, Huang Z, Wu C, Jiang D, Yin L. Preclinical evaluation of IAP0971, a novel immunocytokine that binds specifically to PD1 and fuses IL15/IL15Ralpha complex. Antib Ther. 2022 Nov 17;6(1):38-48. doi: 10.1093/abt/tbac031. eCollection 2023 Jan. PMID 36683766